CLINICAL TRIAL: NCT03557216
Title: Clinical Trial for the Determination of Advanced Colonic Neoplasia Prevalence and the Need for Colonoscopy in Complicated and Uncomplicated Acute Diverticulitis
Brief Title: Acute Diverticulitis and Advanced Colonic Neoplasia. When to Perform Colonoscopy (ADACOLON Study)
Acronym: ADACOLON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADACOLON
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-04

CONDITIONS: Diverticulitis, Colonic; Colonic Neoplasms
Keywords: Diverticulitis; Advanced colonic neoplasm; Colonoscopy
MeSH Terms: conditions — Diverticulitis, Colonic; Colonic Neoplasms; Diverticulitis | interventions — Colonoscopy; Occult Blood

STUDY DESIGN:
Intervention Model Description: Diagnostic clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complicated diverticulitis (Experimental): Patients with complicated diverticulitis diagnosed by computed tomography. Colonoscopy, Fecal immunochemical and occult blood test (FIT) and fecal calprotectin test wil be performed.
  Interventions: Diagnostic Test: Colonoscopy; Diagnostic Test: Fecal immunochemical and occult blood test; Diagnostic Test: Fecal calprotectin test
- Uncomplicated diverticulitis (Experimental): Patients with uncomplicated diverticulitis diagnosed by computed tomography. Colonoscopy, Fecal immunochemical and occult blood test (FIT) and fecal calprotectin test wil be performed.
  Interventions: Diagnostic Test: Colonoscopy; Diagnostic Test: Fecal immunochemical and occult blood test; Diagnostic Test: Fecal calprotectin test

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Anal introduction of a long, flexible, tubular instrument about 1/2-inch in diameter that transmits an image of the lining of the colon so the doctor can examine it for any abnormalities
Diagnostic Test: Fecal immunochemical and occult blood test — A test for fecal occult blood looks for blood in your feces. It can be a sign of a problem in the digestive system, such as a polyp or cancer in the colon.
  Other Names: FIT
Diagnostic Test: Fecal calprotectin test — Calprotectin is a protein released by neutrophils. When there is inflammation in the colon, neutrophils move to the area and release calprotectin, resulting in an increased level in the stool. This test measures the level of calprotectin in stool as a way to detect inflammation and lesions in the colon.

SUMMARY:
This study evaluate the prevalence of advanced colonic neoplasia (ACN) in acute diverticulitis. A sub-analysis of complicated and uncomplicated acute diverticulitis will be made in order to determinate whether there are differences of advanced colonic neoplasia (ANC) prevalence in both groups and to assess if a colonoscopy is necessary.

DETAILED DESCRIPTION:
This is a prospective study that eliminates biases in the selection, design and variability of retrospective studies to reliably assess the global prevalence of advanced colon neoplasia (ACN) and the difference in prevalence among populations with complicated and uncomplicated acute diverticulitis diagnosed by computed tomography. Another objective is to assess the diagnostic prediction of computed tomography to detect ACN in acute diverticulitis. It also aims to assess the safety and quality of colonoscopy in a patient recently diagnosed with acute diverticulitis. Finally, it aims to study whether other diagnostic tools such as the presence of clinical risk symptoms or the performance of fecal biological tests could help in narrowing the indication of colonoscopy in this clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

All patients consecutively diagnosed with acute diverticulitis in the participating hospitals during the study inclusion period will be included. For this purpose, a multidetector computerized tomography confirming the diagnosis of acute diverticulitis must be performed on all patients with initial clinical suspicion.

Exclusion Criteria:

1. Patient refusal to participate in the study.
2. Impossibility of obtaining informed consent by the patient or guardian.
3. Age <18 years and> 85 years
4. Impossibility of performing a diagnostic CT of AD.
5. Intercurrent medical or surgical process with prolonged recovery in time that prevents a colonoscopy before 6 months after the resolution of the episode of acute diverticulitis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Presence of ACN | At the moment of colonoscopy.
  For our study, ANC is all colonic lesions that are advanced adenoma or colorectal cancer. Advanced adenoma is defined as that adenoma with size> 10mm, villous component in> 25% and / or high-grade dysplasia or all serrated lesions> 10mm with or without dysplasia. Colonoscopy is the gold standard for ANC detection.

SECONDARY OUTCOMES:
CT predictive value for ACN detection | At the moment of colonoscopy.
  Assessment of diagnostic prediction of computed tomography to detect ANC in acute diverticulitis.
Clinical symptoms predictive value for ANC detection | At the moment of colonoscopy.
  Assessment of diagnostic prediction of clinical symptoms to detect ANC in acute diverticulitis.
Colonoscopy quality | At the moment of colonoscopy.
  A quality colonoscopy will be considered as a complete colonoscopy, with an adequate preparation according to the Boston scale (score greater than or equal to 2 in all segments) and with resection of all polyps <20mm detected.
Colonoscopy security | 30 days post-colonoscopy.
  Assessment of complications arising from colonoscopy. Mayor complication of colonoscopy is defined as the presence of perforation, hemorrhage, postpolypectomy syndrome, thromboembolic accident, acute myocardial infarction and / or death, and minor complication of colonoscopy for the rest of the events.
FIT predictive value for ANC detection | At the moment of colonoscopy.
  Assessment of diagnostic prediction of FIT to detect ANC in acute diverticulitis.
Fecal calprotectin test predictive value for ANC detection | At the moment of colonoscopy.
  Assessment of diagnostic prediction of fecal calprotectin test to detect ANC in acute diverticulitis.

CONTACTS AND LOCATIONS:
Overall Officials: Agustín Seoane Urgorri, MD, Principal Investigator — Parc de Salut Mar. Hospital del Mar.
Locations (1):
- Parc de Salut Mar. Hospital del Mar., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access will be shared with the principal investigators of all the hospitals that participate in the study

REFERENCES:
- [Background] Stollman N, Smalley W, Hirano I; AGA Institute Clinical Guidelines Committee. American Gastroenterological Association Institute Guideline on the Management of Acute Diverticulitis. Gastroenterology. 2015 Dec;149(7):1944-9. doi: 10.1053/j.gastro.2015.10.003. Epub 2015 Oct 8. No abstract available. PMID 26453777
- [Background] Daniels L, Unlu C, de Wijkerslooth TR, Dekker E, Boermeester MA. Routine colonoscopy after left-sided acute uncomplicated diverticulitis: a systematic review. Gastrointest Endosc. 2014 Mar;79(3):378-89; quiz 498-498.e5. doi: 10.1016/j.gie.2013.11.013. Epub 2014 Jan 14. No abstract available. PMID 24434085
- [Background] Lameris W, van Randen A, Bipat S, Bossuyt PM, Boermeester MA, Stoker J. Graded compression ultrasonography and computed tomography in acute colonic diverticulitis: meta-analysis of test accuracy. Eur Radiol. 2008 Nov;18(11):2498-511. doi: 10.1007/s00330-008-1018-6. Epub 2008 Jun 4. PMID 18523784